CLINICAL TRIAL: NCT00002178
Title: A Phase IIIB Open-Label, Comparative Study to Evaluate Saquinavir Soft Gel Capsule (SGC) Treatment in Combination With Other Antiretrovirals in HIV-1 Infected Antiretroviral-Naive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229J; NR15539
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; RNA, Viral; Dosage Forms; Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Saquinavir; Delavirdine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Saquinavir
Drug: Delavirdine mesylate

SUMMARY:
To determine the proportion of patients whose plasma HIV-1 RNA level falls below the level of detection (< 400 copies/ml) at week 16 and 24 of study therapy. To determine the absolute change in plasma HIV-1 RNA and in absolute CD4 cell count during the 24 weeks of study treatment. To collect safety data on the treatment regimens. To determine the percentage of patients without SQV soft gel capsules resistance-associated mutations at week 24.

DETAILED DESCRIPTION:
Patients are randomized to receive 1 of 3 study regimens: Group A - Saquinavir (SQV) soft gel capsules (sgc) plus 2 reverse transcriptase inhibitors (RTIs), Group B - SQV sgc plus delavirdine plus RTI, and Group C - SQV sgc plus nelfinavir plus RTI (or SQV sgc plus ritonavir plus 2 RTIs).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV RNA >= 5000 copies/ml by Amplicor assay.
* Signed, informed consent from parent or legal guardian for patients less than 18 years old.

Previous treatment with antiretrovirals.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dr Charles Farthing, Los Angeles, California
  - Community Research Initiative, Brookline, Massachusetts

REFERENCES:
- [Background] Cadman J. Roche brings new formulation of saquinavir to FDA. Food and Drug Administration. GMHC Treat Issues. 1997 Apr-May;11(4/5):8. PMID 11364377